CLINICAL TRIAL: NCT06991738
Title: Phase 1/2, Open-Label Study of the Safety, Dosimetry and Efficacy of a 3-Dose Regimen of Escalating Doses of 177Lu-DOTA-EB-TATE in Adult Patients With Metastatic, Radioactive Iodine Non-Responsive Oncocytic (Hurthle-Cell) Thyroid Cancer
Brief Title: 177Lu-DOTA-EB-TATE in Adult Patients With Metastatic, Radioactive Iodine Non-Responsive Oncocytic (Hurthle-Cell) Thyroid Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001532; 001532-DK
Record Dates: First submitted 2025-05-23; First posted 2025-05-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; H(SqrRoot) rthle cell thyroid cancer; 177Lu-DOTA-EB-TATE
MeSH Terms: conditions — Thyroid Neoplasms | interventions — (177)Lu-DOTA-EB-TATE

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 177Lu-DOTA-EB-TATE (Experimental): Open-Label Study of the Safety, Dosimetry and Efficacy of a 3-Dose Regimen of Escalating Doses of 177Lu-DOTA-EB-TATE in Adult Patients with Metastatic, Radioactive Iodine Non-Responsive Oncocytic (Hurthle-Cell) Thyroid Cancer
  Interventions: Drug: 177Lu-DOTA-EB-TATE
- 68Ga-DOTA-TATE PET Scan (Other): The radiopharmaceutical 68Ga-DOTATATE is acquired by the NIH PET department in the Clinical Center. The radiopharmaceutical is synthetized on the day of the study and a premade dose of 5 mCi is administered.
  Interventions: Diagnostic Test: 68Ga-DOTA-TATE PET Scan
- Amino acid infusions (Other): Concomitant administration of an amino acid infusion with the study drug 177Lu-DOTA-EB-TATE is for renal protection.
  Interventions: Other: Amino acid infusions; Drug: 177Lu-DOTA-EB-TATE

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-TATE PET Scan — 68Ga-DOTATATE is administered via intravenous injection of 5 1 mCi in a volume of 3 - 5 ml containing up to 50 micrograms [68Ga] DOTATATE.
  Arms: 68Ga-DOTA-TATE PET Scan
Other: Amino acid infusions — Appropriate amino acid solutions infused for this purpose should have a total lysine and arginine content between 18g and 25g and have an osmolality of <= 1050 mOsmol. Concomitant administration of an amino acid infusion with the study drug 177Lu-DOTA-EB-TATE is for renal protection.
  Arms: Amino acid infusions
Drug: 177Lu-DOTA-EB-TATE — Each single-dose vial contains sodium acetate (24.6 mg/mL), gentisic acid (3.7 mg/mL), L-ascorbate (0.445 mg/mL), DTPA (0.051 mg/mL). 177Lu-DOTA-EB-TATE, is a long-acting radiopharmaceutical for PRRT. It consists of a somatostatin analog peptide (TATE) conjugated with a truncated Evans blue (EB) molecule and the metal chelator 1,4,7,10-tetraazacyclodecane-1,4,7,10-tetraacetic acid (DOTA) with the radioisotope 177Lu stably complexed.
  Arms: 177Lu-DOTA-EB-TATE; Amino acid infusions

SUMMARY:
Background:

Oncocytic (Hurthle cell) thyroid cancer (HTC) is a rare disease with few treatment options. Researchers are developing a radioactive drug that targets a protein that appears in high numbers on HTC cancer cells.

Objective:

To test a radioactive drug (177LuDOTA-EB-TATE) in people with HTC.

Eligibility:

People aged 18 years and older with HTC. The HTC must have failed to respond to conventional radioactive treatment; it must also have spread to other parts of the body.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have imaging scans and a test of their heart function.

177LuDOTA-EB-TATE is infused into a vein. Participants will receive 4 infusions spaced 8 to 12 weeks apart. They will stay in the hospital for 4 to 10 days after each infusion. During and after each infusion, participants will remain in a lead-lined room until their radiation levels go down; this usually takes about 24 hours.

Participants will have 4 to 6 follow-up visits in the weeks after each infusion. Procedures will vary at each visit, but may include more imaging scans; blood and urine tests; and tests of heart function. Participants will have 2 single-photon emission computerized tomography (SPECT) scans. SPECT scans show where the study drug is sticking to tumors or maybe other parts of their body. They will lie on a table while a machine rotates around them. Participants will fill in questionnaires about how their thyroid condition affects their life.

Participants will have follow-ups visits for 5 years after their last study treatment.

DETAILED DESCRIPTION:
Study Description:

The proposed indication is for the treatment of somatostatin receptor-positive radioactive iodine (RAI) non-responsive metastatic oncocytic (Hurthle cell) thyroid (HTC) cancer in adults. We hypothesize that this study will address the following:

* Evaluate if 177Lu-DOTA-EB-TATE is safe and tolerable.
* Analyse early efficacy of 177Lu-DOTA-EB-TATE in metastatic HTC.
* Establish the optimal dose of 177Lu-DOTA-EB-TATE that is characterized by an optimal trade-off between efficacy and toxicity based on Bayesian optimal interval phase I/II time-to-event (TITE-BOIN12).

Objectives:

Primary Objectives:

* To determine the optimal dose of 177Lu-DOTA-EB-TATE that is both safe and shows sufficient efficacy for treatment of metastatic HTC based on TITE-BOIN12 design of phase 1/2 clinical trial.
* To identify the dose-limiting toxicities (DLTs) of escalating doses of 177Lu-DOTA-EB-TATE based on individualized dosimetry.
* To assess the efficacy of 177Lu-DOTA-EB-TATE to improve upon progression-free survival (PFS) at 6 months after the last cycle of the study drug in participants with metastatic RAI-non-responsive HTC.

Secondary Objectives:

* To determine dosimetry in patients following each cycle of 177Lu-DOTA-EB-TATE
* To assess the objective response rate (ORR) and disease control rate (DCR) and association between the specific absorbed dose per lesion of 177Lu-DOTA-EB-TATE.
* To assess the association between the specific absorbed dose per lesion with the tumor response as defined by RECIST 1.1 criteria.
* To assess changes in circulating levels of the tumor marker thyroglobulin (Tg) and anti-Tg antibodies throughout study participation.
* To assess the quality of life (QoL) throughout administration of 177Lu-DOTA-EB-TATE cycles.
* To capture extended safety data by assessing the rate of late adverse events (AEs) and serious adverse events (SAEs).

Endpoints:

Primary Endpoints:

* The primary safety endpoint is a combination of serious adverse events (SAEs), and dose limiting toxicities (DLTs) using CTCAE v5.0. We will also assess the number of participants with treat-related adverse events.
* The primary efficacy endpoint is progression free survival (PFS) at 6 months after the last cycle, where progression is defined by RECIST 1.1 criteria.
* For determination of the optimal dose, each patient will be classified into one of four categories according to the presence or absence of toxicity and efficacy at 8-12 weeks after each cycle and at 6 months after the last cycle.

Secondary Endpoints:

* Radiation-absorbed doses following each cycle of study intervention, normalized to administered activity, including:
* Residence time of 177Lu-DOTA-EB-TATE in liver, spleen, kidneys, whole body and blood pool.
* Specific absorbed dose per organ (Gy/GBq) (using MIRD method as implemented in OLINDA/EXM).
* Cumulative absorbed organ doses (Gy).
* Bone Marrow dose using blood-based method.
* Standardized uptake value (SUV) normalized to lean body mass for maximum (SULmax) in discernible target lesions.
* SULmax in liver, spleen, kidneys, bone marrow and pituitary if visible.
* Tumor response documented as objective response rate (ORR) and disease control rate (DCR) assessed at 24 (+/-2 weeks) and 52 (+/-2 weeks), as well as 2, 3, 4, and 5 years (+/-3 months) after completion of all treatment cycles, as defined by RECIST 1.1 criteria.
* Association between ORR/DCR and tumor absorbed dose using Spearman rank correlation 24 (+/-2 weeks) and 52 (+/-2 weeks), as well as 2, 3, 4, and 5 years (+/-3 months) after last dose of study drug
* Change in thyroglobulin (Tg) and anti-Tg antibodies from baseline to 24 (+/-2 weeks) and 52 (+/-2 weeks) post last dose of the study drug.
* ThyPRO QoL scores at baseline, after each study drug cycle, and at 24 (+/-2 weeks) and 52 (+/-2 weeks) post last dose of the study drug.
* AEs and SAEs at 2, 3, 4, 5 years (+/-3 months) of follow up after last dose of study drug.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged 18 years or older.
* Metastatic RAI-non-responsive and/or RAI-non-avid oncocytic (Hurthle cell) thyroid cancer.
* Progressive disease by RECIST 1.1 criteria, with or without symptoms within the last 12 months. This applies to patients with non-measurable disease by RECIST 1.1 criteria, who will be eligible if they have evidence of progression as defined by the development of new lesions within the last 12 months.
* High expression of SSTR2 in at least one metastatic lesion as documented by 68Ga-DOTATATE PET/CT with SUVmax > SUVmax of the liver consistent with Krenning score of >2 or SUVmax >= 13 based on scan performed within 12 weeks of anticipated enrollment.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnant or breastfeeding.
* NET/PET score of 5 by imaging with 68Ga-DOTATATE PET/CT and 18FDG-PET/CT and defined more than 2 lesions that are SSTR2 negative but 18FDG positive and/or more than 2 lesions that have significantly higher uptake of 18FDG than 68Ga-DOTATATE
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-DOTA-EB-TATE as assessed from medical record.
* Patient weight > 500 lbs. (due to the PET scanner table limit).
* Inability to tolerate at least one modality of diagnostic anatomic imaging, such as CT or MRI.
* Participant has had prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 4 weeks or 4 half-lives (whichever is longer), before the first administration of study drug.
* Previous surgery < 6 weeks prior to the start of participation in this study, or participant has not fully recovered from major surgery, or has suffered significant traumatic injury prior the first dose of study drug or expects to have major surgery during the study period or within 3 months after the last dose of study drug.
* Life expectancy < 6 months as assessed by the treating physician.
* Karnofsky performance status scale < 70%.
* Inability or unwillingness to use adequate contraception prior to study entry and for the duration of study participation, including follow-up (7 months after the last dose of study drug for women and 4 months for men). The adequate contraception consists of intrauterine device, contraceptive implant, hormonal contraception or a double-barrier method. If the patient is status post tubal ligation, status post hysterectomy and/or oophorectomy, or their male partners are status post vasectomy, no additional method of contraception is required.
* Deteriorated renal function, as indicated by a creatinine clearance <60 mL/min calculated by the Cockcroft-Gault Equation. The calculated creatinine clearance can be confirmed by measured creatinine clearance.
* Having only one functional kidney, due to potential nephrotoxicity.
* Patients who have had any prior EBRT dose to either kidney.
* Deteriorated bone marrow function, as indicated by:

  * Hemoglobin (Hb) < 8.0 g/dL
  * White blood cell (WBC) < 2 x10^3/uL
  * Absolute neutrophil count (ANC) < 1.0 x 10^3/L
  * Platelets <100 x 10^3/microL
* Deteriorated liver function, as indicated by one or more of the following:

  * International normalized ratio (INR) > 2.0 for patients that are not on Coumadin
  * Prothrombin time (PTT) > 2 x ULN
  * Total bilirubin > 3 mg/dL
  * Serum albumin < 3.0 g/dL unless prothrombin time is within the normal range
  * Alanine aminotransferase (ALT) > 3 x ULN
  * Aspartate aminotransferase (AST) > 3 x ULN.
* Previous local therapy <4 weeks prior to study entry.
* Extended QTc interval above 480 ms confirmed by 2 ECGs. If the first ECG conducted at the screening visit shows extended QTc interval, potential participants will be asked to repeat an ECG within 30 days to confirm. The second ECG can be conducted at NIH CC or at their outside provider, at their potential expense.
* Toxicities from prior therapies that have not resolved to grade 1 or grade 0 excluding dry mouth syndrome from previous RAI and grade 2 anemia/leukopenia as Hgb>=8 g/dl, WBC >=2 x10^3/uL and ANC >= 1.0 x 10^3 are acceptable for enrollment.
* Active and clinically significant bacterial, fungal, or viral infection, including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness. Radiolabeled ligands may affect the immune response, so people with active and clinically significant infections may become too immunocompromised through participation in this study.
* Known brain metastases and/or carcinomatous meningitis unless these metastases have been treated and stabilized.
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior external beam radiation therapy involving >25% of the bone marrow.
* Unmanageable urinary incontinence rendering the administration of 177Lu-DOTA-EB-TATE unsafe.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence.
* Is unwilling or unable to establish care with a local provider outside of NIH CC
* Inability to understand or unwilling to sign a written informed consent document.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2032-07-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the optimal dose of 177Lu-DOTA-EB-TATE that is both safe and shows sufficient efficacy for treatment of metastatic HTC based on TITE-BOIN12 design of phase 1/2 clinical trial [1, 2]. | 8-12 weeks
To identify the dose-limiting toxicities (DLTs) of escalating doses of 177Lu DOTA EB TATE based on individualized dosimetry. | 8-12 weeks
To assess the efficacy of 177Lu DOTA EB TATE to improve upon progression-free survival (PFS) at 6 months after the last cycle of the study drug in participants with metastatic RAI-non-responsive HTC. | 8-12 weeks

SECONDARY OUTCOMES:
To determine dosimetry in patients following each cycle of 177Lu-DOTA-EB-TATE | 8-12 weeks
To assess the objective response rate (ORR) and disease control rate (DCR) and association between the specific absorbed dose per lesion of 177Lu DOTA EB TATE. | 24 (+/-2 weeks) and 52 (+/-2 weeks), as well as 2, 3, 4, and 5 years (+/-3 months) after last dose of study drug
To assess the association between the specific absorbed dose per lesion with the tumor response as defined by RECIST 1.1 criteria. | 24 (+/-2 weeks) and 52 (+/-2 weeks), as well as 2, 3, 4, and 5 years (+/-3 months) after completion of all treatment cycles
To assess changes in circulating levels of the tumor marker thyroglobulin (Tg) and anti-Tg antibodies throughout study participation. | baseline to 24 (+/-2 weeks) and 52 (+/-2 weeks) post last dose of the study drug
To assess the quality of life (QoL) throughout administration of 177Lu DOTA EB TATE cycles. | at baseline, after each study drug cycle, and at 24 (+/-2 weeks) and 52 (+/-2 weeks) post last dose of the study drug
To capture extended safety data by assessing the rate of late adverse events (AEs) and serious adverse events (SAEs). | 2, 3, 4, 5 years (+/-3 months) of follow up after last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001532-DK.html